CLINICAL TRIAL: NCT06489041
Title: Evaluating the Use of Microarray Pharmacogenetic Testing in Patients With Cancer
Brief Title: Evaluating Microarray Pharmacogenetic Testing in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00114240; LCI-GI-NOS-PGX-003 (Other: Atrium Health)
Record Dates: First submitted 2024-06-17; First posted 2024-07-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenomic Testing (Other): A pharmacogenomic (PGx) microarray (multi-gene) panel will be performed to test for genetic variations in genes related to drug response.
  Interventions: Genetic: Pharmacogenomic Testing with the "Global Diversity Array with Enhanced PGx"

INTERVENTIONS:
Genetic: Pharmacogenomic Testing with the "Global Diversity Array with Enhanced PGx" — Pharmacogenomic (PGx) microarray testing will test for certain pharmcogenes that can guide prescribing of certain cancer treatments and/or supportive care medications.

SUMMARY:
The purpose of this research is to evaluate the impact of a microarray PGx test on prescribing/dosing of drugs and cancer treatments in patients with cancer who are currently eligible for single-gene DPYD testing.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, Phase 2 study. The target population is adults ≥18 years of age who have received or will be receiving standard of care single-gene DPYD (dihydropyrimidine dehydrogenase) PGx testing to help guide dosing for their cancer treatment. Pharmacogenes that will be reported back to participants and providers from the microarray test are expected to take approximately one week and will be evaluated by the PGx team and uploaded to the participant's electronic medical record (EMR). Only clinically actionable results per CPIC and FDA guidelines will be included in the participant report. Participants will be followed on study for approximately 6 months to collect data on the number of drug prescriptions with known drug-gene interactions and potentially actionable results, BPAs fired, and actions taken due to BPAs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* Eligible for standard of care single-gene DPYD testing (i.e., receiving or expected to receive a fluoropyrimidine-based chemotherapy regimen). The potential participant meets inclusion criteria if the standard of care single-gene DPYD test is planned or previously ordered. If previously ordered, consent must occur no later than 60 days from the date the DPYD results were available.
* Willing to provide additional buccal swabs if residual DNA from previous DPYD testing is inadequate for microarray testing.

Exclusion Criteria:

• History of prior allogeneic hematopoietic cell transplantation or liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of potentially actionable results based on pharmacogenomic (PGx) test | Baseline
  A potentially actionable result refers to any genotype or phenotype that is associated with specific drug-gene interactions from the Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines or the FDA's Table of Pharmacogenetic Associations. The number of potentially actionable results is a count variable that represents the total occurrences of such genotypes or phenotypes identified in a participant.

SECONDARY OUTCOMES:
The presence of at least one drug-gene interaction | Baseline, at 3 months and at 6 months after receiving the microarray profiling results
  Drug-gene interactions is defined as an interaction between the medication(s) taken by the subject and the genetic variant(s) the subject possesses based on the PGx test. The presence or absence of such interactions is assessed using the guidelines provided by the Clinical Pharmacogenetics Implementation Consortium (CPIC) or the FDA's Table of Pharmacogenetic Associations. The presence of at least one drug-gene interaction is a binary variable (yes/no).
The presence of at least one PGx best practice advisory (BPA) alert | within 6 months of receiving the microarray profiling results
  BPA alert is fired within the Epic electronic health record (EHR) system for the participant when there is presence of a drug-gene interaction at the time of medication order entry. The presence of at least one PGx best practice advisory (BPA) alert for each participant is a binary variable (yes, no).
Percentage of prescriptions that trigger PGx best practice advisory (BPA) alerts | within 6 months of receiving the microarray profiling results
  Percentage of prescriptions that trigger PGx best practice advisory (BPA) alert among all prescriptions for each participant
Taking actions from PGx best practice advisory alerts | within 6 months of receiving the microarray profiling results
  Taking actions after receiving PGx best practice advisory alerts includes remove or keep drug, order or do not order an e-consult, patient previously tolerated/responded treatment, not appropriate, or other. Taking actions is a binary variable (yes, no).

CONTACTS AND LOCATIONS:
Overall Officials: Jai Patel, PharmD, Principal Investigator — Atrium Health Levine Cancer
Locations (1):
- Atrium Health Levine Cancer, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No